CLINICAL TRIAL: NCT06938256
Title: Comparison of Suboccipital Muscle Inhibition Technique vs Rocabado Exercises on Cervicogenic Headache
Brief Title: Suboccipital Muscle Inhibition Technique vs Rocabado Exercises on Cervicogenic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Affan Iqbal, Assistant Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/02015
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; Suboccipital Muscle Inhibition; Rocabado Exercises
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital Muscle Inhibition (Experimental): Conventional Treatment will be given to this groups, which include heat therapy, cervical muscle stretching, cervical muscle strengthening and manual cervical traction.
  With the patient in the supine position and the eyes closed, the therapist sits behind the subject's head and place the palms of his/her hands beneath it, resting the pads of his/her fingers on the projection of the posterior arch of the atlas. Pressure is exerted upward and toward the therapist. The pressure is maintained for 2 minutes until tissue relaxation had been achieved.
  Patients were assessed for baseline measurements against outcome measures. Patients were given a total of 6 sessions such that 3 sessions per week for the duration of 02 weeks. All patients were reassessed at the end of the baseline and 2nd week of treatment for outcome measures.
  Interventions: Other: Suboccipital Muscle Inhibition
- Rocabado 6x6 Exercises (Experimental): Conventional Treatment will be given to this groups, which include heat therapy, cervical muscle stretching, cervical muscle strengthening and manual cervical traction. Rocabado created 6X6 program for the management of CGH which includes 6 fundamental components, that are-
  Rest position of the tongue:
  The anterior 1/3 of the tongue is placed at the palate with mild pressure, which rests the tongue and jaw musculature and promotes diaphragmatic breathing
  Control of TMJ rotation:
  The jaw is repeatedly opened and closed with the anterior 1/3 of tongue on the palate, which decreases initiating jaw movements (eg protrusive movement in opening, talking or chewing)
  Rhythmic stabilization technique:
  Gentle isometrics in the resting position are performed for jaw opening, closing and lateral deviation to promote muscular relaxation via reciprocal inhibition, which promotes an improved resting position of the jaw through proprioceptive input
  Axial extension of the neck:
  Combined upper cervi
  Interventions: Other: Rocabado 6x6 Exercises

INTERVENTIONS:
Other: Suboccipital Muscle Inhibition — With the patient in the supine position and the eyes closed, the therapist sits behind the subject's head and place the palms of his/her hands beneath it, resting the pads of his/her fingers on the projection of the posterior arch of the atlas. Pressure is exerted upward and toward the therapist. The pressure is maintained for 2 minutes until tissue relaxation had been achieved. The physiotherapist progressively increased the pressure exerted during the 10 minutes of treatment.
  Arms: Suboccipital Muscle Inhibition
Other: Rocabado 6x6 Exercises — Rocabado created 6X6 program for the management of CGH which includes 6 fundamental components, one session under supervision and remaining five sessions by the subject at home.
  These components are:
  * Rest position of the tongue
  * Control of TMJ rotation
  * Rhythmic stabilization technique
  * Stabilized head flexion
  * Axial extension of the neck
  * Shoulder posture
  Arms: Rocabado 6x6 Exercises

SUMMARY:
The purpose of the study is to explore the effectiveness of Suboccipital muscle inhibition technique vs Rocabado exercises on cervicogenic headache. A randomized control trial was conducted at National Institute of Rehabilitation Medicine, Alees Medical Centre Islamabad. The sample size was 40 calculated through G-power 3.1. The participants were divided into two interventional groups each having 20 participants. The study duration was six months. Sampling technique applied was non-probability purposive sampling for recruitment and group randomization using flip coin method. Only 20 to 50 years participants with chronic cervicogenic headache were included in the study. Tools used in this study are Digital Inclinometer, Numeric Pain Rating Scale, Romberg Test and HIT-6 Questionnaire. Data was collected at baseline, and at the end of 2nd week. Data analyzed through SPSS version 27.

DETAILED DESCRIPTION:
Cervicogenic headache is a type of secondary headache that originates from cervical spine dysfunction, particularly involving the upper cervical segments. It is frequently unilateral and is often accompanied by neck stiffness and reduced cervical range of motion. The pain typically radiates from the occipital or suboccipital region to the frontotemporal or retro-orbital areas. It is commonly described as dull and non-throbbing. Cervicogenic Headache constitutes about 14-18% of all chronic headaches, making it a significant concern in musculoskeletal and neurologic clinical practice. The condition often leads to impaired quality of life and mild to moderate disability. Manual therapy and therapeutic exercises are widely used in physiotherapy for management.

The suboccipital region plays a crucial role in postural stability and dural tension regulation due to the presence of myodural bridges between the suboccipital muscles and the dura mater. Dysfunction in these structures can contribute to pain and sensorimotor disturbances in Cervicogenic headache. Suboccipital Muscle Inhibition is a manual technique aimed at relieving tension in these muscles and restoring balance. The technique involves sustained pressure applied to the suboccipital area, helping reduce nociceptive input and improving cerebral spinal fluid flow. Studies have found Suboccipital Muscle Inhibition effective for headache relief and postural improvement. It is recognized for promoting muscular relaxation and decreasing headache intensity. However, more comparative evidence is needed.

Cervical postural alignment plays a significant role in managing musculoskeletal conditions such as cervicogenic headaches. Poor posture, particularly forward head posture, can place excessive strain on the upper cervical spine, contributing to headache symptoms and muscular imbalance. To address these postural deficits, Dr. Mariano Rocabado developed the 6×6 exercise protocol, a structured program aimed at restoring proper cranio-cervical alignment. The protocol includes six exercises performed six times per session, repeated six times daily. These exercises target key elements such as tongue posture, cervical spine control, axial extension, and scapular stabilization. By promoting postural awareness and neuromuscular coordination, the protocol supports improved cervical mechanics. It has been shown to be effective in reducing tension, enhancing movement control, and optimizing cervical posture in individuals with postural dysfunctions.

This study aims to compare the effectiveness of the Suboccipital Muscle Inhibition technique and Rocabado 6×6 exercises in managing cervicogenic headaches. It hypothesizes that both interventions will produce improvements, but one may yield superior outcomes in terms of pain reduction, cervical range of motion, and balance. A randomized clinical trial will be conducted involving 40 participants divided equally into two groups. One group will receive SMI with conventional therapy, and the other will perform Rocabado exercises alongside conventional treatment. The treatment duration will consist of six sessions over two weeks. Both subjective and objective outcome measures will be employed to assess changes.

Participants will be assessed using tools like the Numeric Pain Rating Scale for pain intensity, the Flexion Rotation Test for cervical rotation dysfunction, and the HIT-6 for headache-related disability. Balance will be evaluated using the Romberg test, and cervical Range of motion will be measured with a digital inclinometer. Participants eligible for the study will include adults aged 24-50 years with a history of Cervicogenic headache for over three months. Strict inclusion and exclusion criteria will be followed to ensure sample validity. Patients using pain medication or having contraindications to manual therapy will be excluded. The outcome will be measured before and after the intervention.

Both groups will receive the same conventional treatments such as moist heat, cervical stretching, strengthening exercises, and manual traction. Group A will additionally receive the Suboccipital Muscle Inhibition technique applied for 10 minutes in each session. Group B will perform the Rocabado 6×6 protocol, with one supervised session and five sessions conducted independently each day. All treatments are expected to alleviate pain and restore cervical biomechanics. The hypothesis is that direct dural and postural modulation through Suboccipital Muscle Inhibition may show faster effects, while Rocabado's protocol may offer long-term neuromuscular control benefits. Comparative effectiveness will be analyzed using SPSS software with appropriate statistical tests.

The research is expected to fill the gap in literature regarding the comparative effectiveness of these two distinct but relevant approaches in treating Cervicogenic headache. A clearer understanding of their benefits can guide clinicians in personalizing care for patients with Cervicogenic headache, potentially combining the strengths of both methods. The study also aims to provide cost-effective, non-pharmacological management options that reduce headache recurrence, enhance cervical function, and improve patient quality of life. By establishing evidence-based guidelines, this research may influence future physical therapy protocols and headache rehabilitation strategies, ensuring optimized outcomes for Cervicogenic headache sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of chronic CGH (>3 months)

  * CGH pain intensity between 3 and 8 on NPRS
  * Participants who had a unilateral headache that do not shift side (ipsilateral neck pain/stiffness)
  * Pain at least once a week in the previous three months, chronic, episodic, and duration one hour to weeks (non-throbbing pain starts in the neck).
  * CGH due to cervical spine dysfunction
  * Neck pain followed by headache
  * Patients with neck stiffness and movement restriction were included.
  * Flexion Rotation Test results that are positive with a restriction of more than 10 degrees.

Exclusion Criteria:

* Participants with other types of headache migraine, sinus, tumor, neural, or temporomandibular joint issues)
* Cervicogenic headache patients with mixed headache or any diagnosed serious pathology of alar ligament and vertebra basilar artery insufficiency
* Any contraindications to manual and manipulative therapy (fracture, instability, osteoporosis, arthropathy, or neural symptoms)
* Using analgesics or corticosteroids
* Metastasis
* Cardiac conditions (stroke, hypertension, or syncope)
* Neurological conditions (radiculopathy, myelopathy, or disc problems)
* Spinal cord problem
* Previous brain and spinal cord surgery
* Occlusal splints or any surgery in Temporomandibular joint area.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Numeric Pain Rating Scale | 2nd week
  Change from baseline the NPRS score and 2nd week. NPRS is the ideal to measure pain intensity of pain. It has scale of 0-10 ("0" = no pain and "10" = worst imaginable pain).

SECONDARY OUTCOMES:
Changes from baseline in cervical range of motion | 2nd week
  ROM Cervical Spine (Flexion) Changes from the Baseline ROM range of Motion of Cervical spine flexion was taken with the Help of Digital Inclinometer ROM Cervical Spine (extension) Changes from the Baseline ROM range of Motion of Cervical spine extension was taken with the Help of Digital Inclinometer ROM Cervical Spine (Right side flexion) Changes from the Baseline ROM range of Motion of Cervical spine right side flexion was taken with the Help of Digital Inclinometer ROM Cervical Spine (left side Flexion) Changes from the Baseline ROM range of Motion of Cervical spine left side flexion was taken with the Help of Digital Inclinometer ROM Cervical Spine (right rotation) Changes from the Baseline ROM range of Motion of Cervical spine right rotation was taken with the Help of Digital Inclinometer ROM Cervical Spine (left rotation) Changes from the Baseline ROM range of Motion of Cervical spine left rotation was taken with the help of Digital Inclinometer.
Changes from baseline in HIT-6 Questionnaire | 2nd week
  Changes from baseline in HIT-6 Questionnaire were taken.The HIT-6, a 6-item questionnaire, designed to measure patient's severity and frequency of headache and impact on daily life.
Changes from baseline in Romerg's Test | 2nd week
  The changes from baseline were taken with the help of Romberg test which is a simple clinical assessment used to evaluate a person's balance and proprioception. The patient stands with feet together, arms at the sides, first with eyes open, then closed. A positive test-marked by increased swaying or loss of balance with eyes closed-indicates impaired proprioceptive or vestibular function.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Rehabilitation and Medicine, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No